CLINICAL TRIAL: NCT00004895
Title: Octreotide for Palliation of Inoperable Bowel Obstruction: A Phase II Study
Brief Title: Octreotide as Palliative Therapy for Cancer-Related Bowel Obstruction That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: NU 97X1; NU-97X1; NCI-G00-1685
Record Dates: First submitted 2000-03-07; First posted 2003-05-09 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Colorectal Cancer; Constipation, Impaction, and Bowel Obstruction; Extrahepatic Bile Duct Cancer; Gastric Cancer; Gastrointestinal Stromal Tumor; Nausea and Vomiting; Ovarian Cancer; Pancreatic Cancer; Peritoneal Cavity Cancer; Small Intestine Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent pancreatic cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; small intestine adenocarcinoma; small intestine lymphoma; small intestine leiomyosarcoma; localized extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; recurrent small intestine cancer; constipation, impaction, and bowel obstruction; peritoneal cavity cancer; nausea and vomiting; gastrointestinal stromal tumor
MeSH Terms: conditions — Colorectal Neoplasms; Constipation; Intestinal Obstruction; Bile Duct Neoplasms; Stomach Neoplasms; Gastrointestinal Stromal Tumors; Nausea; Vomiting; Ovarian Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: octreotide acetate

SUMMARY:
RATIONALE: Palliative therapy with octreotide may help patients who have bowel obstruction that cannot be removed by surgery to live longer and more comfortably.

PURPOSE: Phase II trial to study the effectiveness of octreotide as palliative therapy in treating patients who have cancer-related bowel obstruction that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effectiveness of octreotide in the palliation of bowel obstruction secondary to cancer.
* Characterize the dose and tolerability of octreotide in this patient population.

OUTLINE: Patients receive octreotide subcutaneously or IV over 24 hours on days 2-5.

Patients who respond well to study may continue octreotide for palliative effects.

PROJECTED ACCRUAL: A total of 9-25 patients will be accrued for this study over 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Inoperable bowel obstruction secondary to cancer OR
* Metastatic or primary abdominal cancer
* Patient presents with vomiting
* Percutaneous gastrostomy tube allowed

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-4

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No documented hypersensitivity to octreotide
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior chemotherapy allowed

Endocrine therapy:

* Concurrent steroids allowed

Radiotherapy:

* Prior radiotherapy allowed

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Cameron Muir, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States